CLINICAL TRIAL: NCT04018326
Title: Causes and Clinical Impact of Loss to Follow-up in Patients With Proliferative Diabetic Retinopathy
Brief Title: Loss to Follow-up in PDR Patients
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Abdelazeem, Associate Professor of Ophthalmology, Assiut University
Other Study IDs: 17300291
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Diabetic Retinopathy
Keywords: loss to follow-up; proliferative diabetic retinopathy; diabetic retinopathy; panretinal photocoagulation; intravitreal injections
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Compliant patients: The compliant patient was defined as a patient who did not miss any follow-up visit until the end of the study period.
- Loss to follow-up (LTFU): LTFU was defined as missing any follow-up visit for any interval exceeding 6 months provided that patients eventually resumed care before the end of the study period (time zero was defined as the date of the missed follow-up visit).

SUMMARY:
This study determined the clinical impact and causes of loss to follow-up (LTFU) from the patients' perspective in individuals with proliferative diabetic retinopathy (PDR) who received panretinal photocoagulation (PRP) and/or intravitreal injections (IVIs) of anti-vascular endothelial growth factor (VEGF).

This prospective cohort study included 467 patients with PDR who received PRP and/or IVIs of anti-VEGF between May 2013 and June 2018. LTFU was defined as missing any follow-up visit for any interval exceeding 6 months, provided that patients eventually resumed care. Main outcome measures include rates and causes of LTFU.

ELIGIBILITY:
Inclusion Criteria:

* included treatment-naïve patients who had developed PDR in one eye with a best corrected visual acuity (BCVA) ranging from 20/22 to 20/69, as determined by the Snellen equivalent. Patients were allocated to receive PRP, IVIs of anti-VEGF, or a combination of both procedures.

Exclusion Criteria:

1. patients receiving follow-up ophthalmic care for their PDR with or without interventions at any other medical care provider during the observation period, as declared by the patients at any follow up visit.
2. patients LTFU who did not resume follow-up until the end of the observation period.
3. patients needing PPV at first presentation or having additional retinal pathology. 4) patients receiving their treatment procedure during December 2017 or having vitreous hemorrhage that failed to clear up by June 2018 but still ineligible candidates for PPV.

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients who had developed PDR in one eye. Patients were allocated to receive PRP, IVIs of anti-VEGF, or a combination of both procedures.
Sampling Method: Non-Probability Sample
Enrollment: 467 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-12-25 (Actual)

PRIMARY OUTCOMES:
Final BCVA | "through study completion, an average of 1 year",
  logMAR BCVA at final follow up (Snellen equivalent)
Final UCVA | "through study completion, an average of 1 year",
  Final logMAR UCVA (Snellen equivalent)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdelmotaal H, Ibrahim W, Sharaf M, Abdelazeem K. Causes and Clinical Impact of Loss to Follow-Up in Patients with Proliferative Diabetic Retinopathy. J Ophthalmol. 2020 Feb 8;2020:7691724. doi: 10.1155/2020/7691724. eCollection 2020. PMID 32089871

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-02-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT04018326/Prot_SAP_000.pdf